CLINICAL TRIAL: NCT06419101
Title: Cohort Study on Biomarkers of Cognitive Disorders in China
Brief Title: Exploring the Diagnostic Biomarkers of Cognitive Disorders in China
Status: Recruiting | Type: Observational
Sponsor: Cuibai Wei，Clinical Professor (Other)
Collaborators: First Hospital of Shijiazhuang City (Other); Chongqing Medical University (Other); Tianjin Huanhu Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Sponsor-Investigator, Cuibai Wei，Clinical Professor, Xuanwu Hospital, Capital Medical University, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: KS2024051
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Biomarkers; Dementia
Keywords: dementia; diagnostic biomarkers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, CSF, urine, faeces, saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dementia progression: dementia-P (Compared with the baseline, MMSE score declined ≥ 4 points per year)
- dementia stabilization: dementia-S (Compared with the baseline, MMSE score decreased < 4 points per year）

SUMMARY:
Dementia is a syndrome characterized by progressive global cognitive impairment that impairs occupational, family, or social functioning. It detrimentally affects personal health and quality of life, imposing significant medical economy, social and psychological burden on the countries and the patients' family. The internationally renowned dementia cohort includes the DIAN that focused on genetics studies, the ADNI cohort featuring imaging and the FINGERS cohort focused on risk factor intervention, etc. Establishing standardized and shared longitudinal follow-up dementia cohorts and clinical database is an essential challenge for constructing dementia cohort in China. Moreover, there is a lack of large-scale prospective longitudinal follow-up cohorts within the Chinese population that cover subjective cognitive decline (SCD) to explore biomarkers with diagnostic and early warning value for different kinds of dementia and pre-dementia stages. The study will rely on the dementia cohort based on Chinese population to explore the biological phenotype characteristics of the pre-dementia stage and different dementia subtypes, and observe the dynamic change rules of the dementia cohort vertically, so as to foster early intervention and improve prognosis for individuals with dementia.

DETAILED DESCRIPTION:
The 3000 patients with pre-dementia stage and different dementia subtypes will be enrolled in this study, and data will be collected in the baseline including demographics, clinical symptoms, assessment of neuropsychology, neuroimaging, neuroelectrophysiology, blood samples, cerebrospinal fluid, etc. The changes of these data were dynamically observed through an annual follow-up. According to the neuropsychological evaluation results of follow-up, the subjects were divided into dementia progression (dementia-P) and dementia stabilization (dementia-S). Difference in clinical phenotype, neuropsychology, electrophysiology, neuroimaging, and body fluid multi-omics indicators between the two subtypes were compared and analyzed. The neuropsychological testes in patients with dementia included some neuropsychological scales such as, Clinical Dementia Rating (CDR), Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), etc. Multi-model neuroimaging evaluation screen the candidate neuroimaging markers, including structure and functional brain magnetic resonance imaging (MRI), Diffusion tensor image (DTI), 18 F-2-fluro-D-deoxy-glucose-positron emission tomography (18F-FDG-PET)，Amyloid-PET and tau-PET. To exploring neuroelectrophysiology biomarkers collect the data on polysomnography, resting state electroencephalogram, and evoked potentials (P1, N1, P2, N2, etc.). ELISA, SIMOA and other analytical methods were used to detect the contents related to dementia progression in the blood, cerebrospinal fluid, urine, saliva and feces. Multi-dimensional screening and identifying biomarkers of disease diagnosis and progression in all stages, from subjective cognitive impairment to mild cognitive impairment to dementia, in line with the characteristics of the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥40 and ≤90years;
* Chief complaint or others describe a cognitive decline;
* Ability to communicate in Chinese;
* The patients and their families were informed and signed the informed consent.

Exclusion Criteria:

* MMSE<10;
* There are other neurological diseases that can cause brain dysfunction (such as depression, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, traumatic brain injury, normal intracranial pressure hydrocephalus, etc.);
* There are other systemic diseases that can cause cognitive impairment (such as hepatic insufficiency, renal insufficiency, Thyroid dysfunction, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
* Suffering from a disease that cannot cooperate with the completion of cognitive examination;
* There are contraindications to nuclear magnetic resonance;
* There is mental and neurodevelopmental delay;
* Refuse to draw blood;
* Refuse to sign the informed consent.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project will enroll about 3000 patients with dementia, who meet the inclusion and exclusion criteria, including subjective cognitive decline (SCD), MCI, AD, frontotemporal dementia (FTD), dementia with Lewy bodies (DLB), etc.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2034-05-10 (Estimated); Study Completion 2035-05-10 (Estimated)

PRIMARY OUTCOMES:
Rate of change in global cognition as measured by Clinical Dementia Rating (CDR). | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales CDR. CDR, a multidimensional scale for dementia severity, which scored 0-3, with higher scores indicating worse functioning.

SECONDARY OUTCOMES:
Rate of change in global cognition as measured by Mini-Mental State Examination (MMSE) | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales MMSE. MMSE scores range from 0-30, with higher scores representing better cognitive function.
Rate of change in global cognition as measured by Montreal Cognitive Assessment (MoCA) | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales MoCA. MoCA scores range from 0-30, with higher scores representing better cognitive function.
Rate of change in the severity of cognitive impairment as assessed by Alzheimer's Disease Assessment Scale-Cognitive section (ADAS-cog). | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales ADAS-cog. ADAS-cog scores range from 0-70, with higher scores indicating better global cognitive function.
Rate of change in memory function as assessed by World Health Organization-University of California, Los Angeles, auditory verbal learning test (WHO-UCLA AVLT). | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales like WHO-UCLA AVLT. WHO-UCLA AVLT scores depend on the number of correct words, which ranges from 0-15, with higher scores representing better memory function.
Rate of change in language function as assessed by Boston Naming Test (BNT). | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales like BNT. BNT scores range from 0-30, with higher scores representing better language function.
Rate of change in psychobehavioral symptoms as assessed by Neuropsychiatric Inventory (NPI). | 10 years
  Assess statistically significant difference in score between dementia-P and dementia-S using the neuropsychological scales like NPI. Patient assessment grading scores range from 0-144 in NPI, and caregivers distress grading scores range from 0-60, with 0 representing the best.
Rate of change in activities of daily living as assessed by Alzheimer's Disease Cooperative Study-Activity of Daily Living (ADCS-ADL). | 10 years
  Assess statistically significant difference between in score dementia-P and dementia-S using the neuropsychological scales like ADCS-ADL. ADCS-ADL scores range from 0-54, with higher scores indicating better completion ability.

CONTACTS AND LOCATIONS:
Overall Officials: Cuibai Wei, Principal Investigator — Xuan Wu Hospital of Capital Medical University, Beijing, China, 100053
Locations (1):
- Capital Medical University Xuanwu Hospital, Beijing, China